CLINICAL TRIAL: NCT05680077
Title: Methylation Detection of KCNA3 and OTOP2 Genes in Plasma for the Auxiliary Diagnosis of Esophageal Cancer/Precancerous Lesions: a Clinical Trial
Brief Title: KCNA3 and OTOP2 Gene Methylation Combined Detection Kit (Fluorescent PCR Method)
Status: Completed | Type: Observational
Sponsor: Wuhan Ammunition Life-tech Co., Ltd (Industry)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AD10
Record Dates: First submitted 2022-12-08; First posted 2023-01-11 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal carcinoma; Esophageal high-grade intraepithelial neoplasia; methylation; Fluorescent PCR
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — human blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: Esophageal carcinoma and high-grade intraepithelial neoplasia patients.
  Interventions: Diagnostic Test: KCNA3 and OTOP2 Gene Methylation Combined Detection Kit (Fluorescent PCR Method)
- Negative group: Patients with other digestive malignancies (including gastric cancer, colorectal cancer, liver cancer, pancreatic cancer,Cholangiocarcinoma, etc.) and patients with non-digestive malignant tumors (including thyroid cancer, lung squamous cell carcinoma, cervix Cancer, endometrial cancer, breast cancer, prostate cancer, etc.), Patients with benign digestive disorders (including esophagitis, gastritis, enteritis, appendicitis, gastric polyps, colorectal polyps, etc.).
  Interventions: Diagnostic Test: KCNA3 and OTOP2 Gene Methylation Combined Detection Kit (Fluorescent PCR Method)

INTERVENTIONS:
Diagnostic Test: KCNA3 and OTOP2 Gene Methylation Combined Detection Kit (Fluorescent PCR Method) — Blood samples from participants in both groups were collected and methylation tests were performed according to the kit instructions.

SUMMARY:
The goal of this observational study is to test the clinical efficacy of "KCNA3 and OTOP2 gene methylation combined detection kit (fluorescence PCR method)"in esophageal cancer and high-grade esophageal neoplasia auxiliary diagnosis.The main questions it aims to answer are:

1. How consistent are the test results of the kit with the clinical reference diagnostic criteria?
2. Sanger sequencing can visually show whether each sample contains methylation sites, so in this clinical trial, the kit results were compared with Sanger sequencing results to analyze the reagent's accuracy in detecting KCNA3 and OTOP2 gene methylation.

Each participant is required to provide no less than 10 ml of blood to complete the kit test.

DETAILED DESCRIPTION:
Esophageal carcinoma is caused by abnormal hyperplasia of the squamous or glandular epithelium, the main pathological types are squamous cell carcinoma and adenocarcinoma. Globally, esophageal cancer has the seventh highest incidence and the sixth leading cause of cancer death. Statistics showed that in 2020, there were 604,000 new cases of esophageal cancer and 54.4 deaths.

The 5-year survival rates were significantly different in esophageal carcinomas of different stages, for example, it's 84.9% for stage Ia, 70.9% for stage Ib, 56.2% for stage IIa, 43.3% for stage IIb, 37.9% for stage IIIa, 23.3% for stage IIIb, 12.9% for stage IIIc and 3.4% for stage IV. Therefore, early diagnosis and treatment is most effective strategy to reduce the incidence and mortality of esophageal cancer.

Endoscopy and pathological biopsy are currently the "golden standard" for diagnosing esophageal cancer, however, limited by medical resources, tolerance and other issues, population screening by endoscopy is not cost-effective and applicable. There is no recognized and effective serologic marker for the detection of early esophageal carcinoma and precancerous lesions, the effect of multiple serological markers combined detection is better than that of single markers, and the accuracy were 74%~85% , but it is still suboptimal.

Methylation of the tumor suppressor gene promoter region CpG island is the most common change during tumorgenesis, studies showed that methylation events could occur at the early stages of esophageal cancer.

Circulating tumor DNA (ctDNA) is derived from DNA fragments produced by apoptosis, necrosis or secretion of tumor cells, which is a part of circulating free (cfDNA). CtDNA contains the same gene defects as its source tumor DNA, such as point mutation, rearrangement, amplification, microsatellite change, epigenetic modification, etc.

KCNA3 is a member of the protein family that encodes potassium channels and mainly affects cell viscosity. OTOP2 is a member of the protein family encoding proton transport channels, some studies have shown that the methylation levels of two genes in esophageal cancer tissues were significantly higher than that in adjacent tissues, and they can be used as a potential marker for the diagnosis of esophageal cancer.

This kit is based on real-time fluorescence PCR technology to achieve the qualitative detection of KCNA3 and OTOP2 methylation in plasma samples. Before PCR amplification, cfDNA was transformed by bisulfite and ACTB (β-Actin) gene is used us the internal reference.

ELIGIBILITY:
Inclusion Criteria:

1. esophageal carcinoma patients confirmed or highly suspected by endoscopy, imaging examination or pathological biopsy, and high-grade intraepithelial neoplasia of the esophagus patients mainly enrolled from individuals who planned to undergo radical esophagectomy of esophageal cancer, endoscopic submucosal dissection or primary chemoradiotherapy.
2. patients with benign diseases of digestive system who have undergone endoscopy (including esophagitis, gastritis, enteritis, appendicitis, gastric polyps, colorectal polyps, etc.).
3. Untreated patients with other digestive system malignancies (including gastric cancer, colorectal cancer, liver cancer, pancreatic cancer, bile duct cancer, etc.) and patients with non-digestive system malignancies (including thyroid cancer, lung squamous cell carcinoma, cervical cancer, endometrial cancer, breast cancer, prostate cancer, etc.) confirmed by clinical reference diagnostic criteria.

Exclusion Criteria:

1. patients who have received anti-tumor therapy such as radiotherapy/chemotherapy;
2. Esophageal carcinoma and high-grade intraepithelial neoplasia patients who were also suffering from other malignant tumors;
3. Samples not kept as required or samples of hemolysis;
4. The sample volume fails to meet the detection requirements;
5. Esophageal carcinoma patients with distant metastasis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Esophageal cancer patients, number ≥ 300, containing different TNM stages.
  2. Esophageal high-grade intraepithelial neoplasis patients, number ≥70.
  3. Patients with benign diseases of digestive system including esophagitis, gastritis, enteritis, appendicitis, gastric polyps, colorectal polyps, etc. , number ≥200.
  4. Patients with other digestive system malignancies (including gastric cancer, colorectal cancer, liver cancer, pancreatic cancer, bile duct cancer, etc.) and patients with non-digestive system malignancies (including thyroid cancer, lung squamous cell carcinoma, cervical cancer, endometrial cancer, breast cancer, prostate cancer, etc.)， number ≥350.
  5. All the enrolled participants should be ≥1000.
Sampling Method: Probability Sample
Enrollment: 1116 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
validity | Immediately after the procedure
  In this study, validity indicates the consistency of methylation test with the golden diagnostic standards, including sensitivity and specificity. Sensitivity indicates the proportion of methylation-positive samples in esophageal cancer/high-grade neoplasia samples. Specificity indicates the proportion of methylation-negative samples in non-esophageal cancer/high-grade neoplasia.

SECONDARY OUTCOMES:
reliability | Immediately after the procedure
  In this study, the reliability evaluation included two indicators, namely the agreement rate of methylation detection with Sanger sequencing, and the Kappa value of the two methods

CONTACTS AND LOCATIONS:
Overall Officials: Luowei Wang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- The First Affiliated Hospital of Naval Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Confidential information of the individual participant will be retained by investigators and clinical trial institutions, any personal information of subjects will not be disclosed in reports, publications, etc.
  Direct access to source data and and files is only allowed for the purpose of monitoring, auditing or inspection, without revealing the subject's privacy.
  The medical products administration may inspect the basic documents of clinical trials of medical devices in order to confirm the authenticity and the integrity of the collected data.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Wang GQ, Abnet CC, Shen Q, Lewin KJ, Sun XD, Roth MJ, Qiao YL, Mark SD, Dong ZW, Taylor PR, Dawsey SM. Histological precursors of oesophageal squamous cell carcinoma: results from a 13 year prospective follow up study in a high risk population. Gut. 2005 Feb;54(2):187-92. doi: 10.1136/gut.2004.046631. PMID 15647178
- [Background] di Pietro M, Canto MI, Fitzgerald RC. Endoscopic Management of Early Adenocarcinoma and Squamous Cell Carcinoma of the Esophagus: Screening, Diagnosis, and Therapy. Gastroenterology. 2018 Jan;154(2):421-436. doi: 10.1053/j.gastro.2017.07.041. Epub 2017 Aug 2. PMID 28778650
- [Background] Wang J, Wu N, Zheng QF, Yan S, Lv C, Li SL, Yang Y. Evaluation of the 7th edition of the TNM classification in patients with resected esophageal squamous cell carcinoma. World J Gastroenterol. 2014 Dec 28;20(48):18397-403. doi: 10.3748/wjg.v20.i48.18397. PMID 25561808
- [Background] Talukdar FR, Soares Lima SC, Khoueiry R, Laskar RS, Cuenin C, Sorroche BP, Boisson AC, Abedi-Ardekani B, Carreira C, Menya D, Dzamalala CP, Assefa M, Aseffa A, Miranda-Goncalves V, Jeronimo C, Henrique RM, Shakeri R, Malekzadeh R, Gasmelseed N, Ellaithi M, Gangane N, Middleton DRS, Le Calvez-Kelm F, Ghantous A, Roux ML, Schuz J, McCormack V, Parker MI, Pinto LFR, Herceg Z. Genome-Wide DNA Methylation Profiling of Esophageal Squamous Cell Carcinoma from Global High-Incidence Regions Identifies Crucial Genes and Potential Cancer Markers. Cancer Res. 2021 May 15;81(10):2612-2624. doi: 10.1158/0008-5472.CAN-20-3445. Epub 2021 Mar 19. PMID 33741694
- [Background] Qin Y, Wu CW, Taylor WR, Sawas T, Burger KN, Mahoney DW, Sun Z, Yab TC, Lidgard GP, Allawi HT, Buttar NS, Smyrk TC, Iyer PG, Katzka DA, Ahlquist DA, Kisiel JB. Discovery, Validation, and Application of Novel Methylated DNA Markers for Detection of Esophageal Cancer in Plasma. Clin Cancer Res. 2019 Dec 15;25(24):7396-7404. doi: 10.1158/1078-0432.CCR-19-0740. Epub 2019 Sep 16. PMID 31527170
- [Background] Cao W, Lee H, Wu W, Zaman A, McCorkle S, Yan M, Chen J, Xing Q, Sinnott-Armstrong N, Xu H, Sailani MR, Tang W, Cui Y, Liu J, Guan H, Lv P, Sun X, Sun L, Han P, Lou Y, Chang J, Wang J, Gao Y, Guo J, Schenk G, Shain AH, Biddle FG, Collisson E, Snyder M, Bivona TG. Multi-faceted epigenetic dysregulation of gene expression promotes esophageal squamous cell carcinoma. Nat Commun. 2020 Jul 22;11(1):3675. doi: 10.1038/s41467-020-17227-z. PMID 32699215
- [Background] Tu YH, Cooper AJ, Teng B, Chang RB, Artiga DJ, Turner HN, Mulhall EM, Ye W, Smith AD, Liman ER. An evolutionarily conserved gene family encodes proton-selective ion channels. Science. 2018 Mar 2;359(6379):1047-1050. doi: 10.1126/science.aao3264. Epub 2018 Jan 25. PMID 29371428